CLINICAL TRIAL: NCT06434584
Title: Explainable Insulin Decision-making System to Assist Physicians in Diabetes Management
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20240218043800077
Record Dates: First submitted 2024-05-09; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- senior doctor group
  Interventions: Other: without AI assistance; Other: with AI dosage assistance; Other: with explainable AI assistance; Other: with faulty explainable AI assistance
- junior doctor group
  Interventions: Other: without AI assistance; Other: with AI dosage assistance; Other: with explainable AI assistance; Other: with faulty explainable AI assistance

INTERVENTIONS:
Other: without AI assistance — provide insulin dosage and confidence score without AI assistance
Other: with AI dosage assistance — provide insulin dosage and confidence score with AI dosage assistance
Other: with explainable AI assistance — provide insulin dosage and confidence score with explainable AI assistance
Other: with faulty explainable AI assistance — provide insulin dosage and confidence score with faulty explainable AI assistance

SUMMARY:
The investigators plan to conduct a multi-case, multi-reader observational study with the primary objective of exploring the effects of an interpretable insulin-assisted decision-making system on physicians' (1) decision accuracy and (2) decision confidence.

ELIGIBILITY:
Case:

Inclusion Criteria:

* Patients with T2DM who were admitted to Zhongshan Hospital of Fudan University from 2022.12 to 2023.3.
* Insulin regimen is one of the following: a. Basal regimen: once a day subcutaneous injection of long-acting or ultra-long-acting insulin; b. Premixed regimen: two/three times a day subcutaneous injection of premixed insulin; c. Basal mealtime regimen: three times a day before meals subcutaneous injection of short-acting or rapid-acting insulin, plus once a day injection of long-acting or ultra-long-acting insulin.

Exclusion Criteria:

- Cases will be excluded if there is insufficient information for a valid assessment (missing data on insulin or blood glucose >40%).

Doctor

Inclusion Criteria:

licensed medical practitioner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: include 40 patient cases and 8 doctors (4 senior and 4 junior)
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-12-10 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Doctors' decision-making accuracy | up to 2 months
  The investigators used MAE and clinical agreement to quantitatively assess the accuracy of clinician-recommended insulin doses.
  1. Mean Absolute Error (MAE) represents the error between the clinician-recommended value and the expert-recommended value (gold standard).
  2. Clinical agreement: Clinical agreement is calculated as the proportion of clinically consistent insulin doses (clinician-given adjustments in the same direction as the expert's protocol and within 20% of the dose difference) to the total insulin dose.
Doctors' decision-making confidence | up to 2 months
  Clinicians' confidence in decision-making was assessed using a 10-point Likert scale from 1 (not at all confident) to 10 (completely confident).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Li, Professor, Study Chair — Fudan University
Locations (1):
- Xiaoying Li, Shanghai, Shanghai Municipality, China